CLINICAL TRIAL: NCT04594707
Title: A Phase III Open-label Extension Study to Evaluate Long-term Safety and Efficacy of PRM-151 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Evaluate Long Term Safety and Efficacy of Recombinant Human Pentraxin-2 (rhPTX-2; PRM-151) in Participants With Idiopathic Pulmonary Fibrosis
Acronym: STARSCAPE-OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by Sponsor as the futility analysis outcome indicated that the study was unlikely to meet the predefined primary objective of the study. No new safety concerns were identified.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA42294; 2020-001429-30 (EudraCT Number)
Record Dates: First submitted 2020-10-15; First posted 2020-10-20 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — PRM-151

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zinpentraxin Alfa (Experimental): Corhort A: Participants entering, following participation in study PRM-151-202.
  Cohort B: Participants entering, following participation in study WA42293.
  Interventions: Drug: PRM-151 (Zinpentraxin Alfa)

INTERVENTIONS:
Drug: PRM-151 (Zinpentraxin Alfa) — Cohort A: Participants will receive three loading doses of open-label PRM-151 on days 1, 3, and 5, then one infusion every 4 weeks (Q4W). 10 mg/kg of PRM 151 will be administered by intravenous (IV) infusion over 60 minutes on days 1, 3, and 5, then one infusion every 4 weeks.
  Cohort B: Participants previously randomized to the placebo in WA42293 will receive study medication in the three loading doses on days 1, 3 and 5 in a blinded fashion. All three doses will contain PRM-151. Participants previously randomized to the treatment arm in WA42293 will receive study medication in the three loading doses on days 1, 3 and 5 in a blinded fashion. One of the three doses will contain PRM-151, whereas two doses will contain placebo.
  Other Names: Zinpentraxin Alfa

SUMMARY:
This study will evaulate the long-term safety, efficacy and pharmacokinetics (PK) of recombinant human pentraxin-2 (rhPTX-2; PRM-151) zinpentraxin alfa, administered by intravenous (IV) infusion to participants with idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
This study is being conducted for the treatment of eligible participants who have taken part in Study PRM-151-202 and received the open-label study drug or completed the Phase III Study WA42293 with PRM-151. Participants who have discontinued treatment from or have completed Study WA42293 and do not want to receive PRM-151 in this study, will be invited to enroll in survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Taken part in either of the prior PRM-151 studies: PRM-151-202 or WA42293.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.

Exclusion Criteria:

* Acute respiratory or systemic bacterial, viral, or fungal infection at the first visit of the OLE, or within 2 weeks of the first visit for patients joining Cohort A (from Study PRM-151-202).
* History of smoking within 3 months prior to the first visit in the OLE.
* History of alcohol or substance use disorder within 2 years prior to the first visit of the OLE or known or suspected active alcohol or substance-use disorder.
* History of severe allergic reaction or anaphylactic reaction to PRM-151.
* Clinically significant abnormality on ECG during eligibility assessment that, in the opinion of the investigator, may pose an additional risk in administering study drug to the participant.
* Prolonged corrected QT interval > 450 ms (for men) or > 470 ms (for women) based on the Fridericia correction formula.
* Clinically significant laboratory test abnormalities (hematology, serumchemistry, and urinalysis) that, in the opinion of the investigator, may pose an additional risk in administering study drug to the participant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (248):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis, Sacramento, California
  - Inst. of Healthcare Assessment, Inc., San Diego, California
  - UCSF Medical Center, San Francisco, California
  - National Jewish Health Medical Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Meris Clinical Research, Brandon, Florida
  - Florida Lung, Asthma and Sleep Specialists (FLASS) - Celebration, Celebration, Florida
  - Advanced Pulmonary & Sleep Research Institute of Florida, Daytona Beach, Florida
  - University of Florida Health Pulmonology - Jacksonville, Jacksonville, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Sarasota County Public Hospital, Sarasota, Florida
  - Renstar Medical Research, Wesley Chapel, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - University of Iowa Hospitals and Clinics; Investigational Drug Services, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Lung Research Center, Chesterfield, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Lenox Hill Hospital, New York, New York
  - Pulmonix Research, Greensboro, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson University Physicians (JUP) - Jefferson Pulmonary, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Lowcountry Lung and Critical Care, North Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - University Of Utah Hosp & Clin; Investigational Pharmacy, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (10):
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Respirar (Centro Medico Dra. De Salvo), Ciudad Autonoma Buenos Aires
  - Instituto de Medicina Respiratoria, IMeR; Clinic/Outpatient Facility, Córdoba
  - Hospital Universitario Austral, Derqui-Pilar
  - Centro Medico de Enfermedades Respiratorias (CEMER), Florida, Buenos Aires
  - Centro de estudios respiratorios, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza, Mendoza City
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Cairns Base Hospital; Cancer Care Centre, Cairns, Queensland
  - Lung Research Queensland, Nundah, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre; Medicine, Melbourne, Victoria
  - The Alfred Hospital, Prahan, Victoria
- Belgium (5):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc; Pharmacy, Brussels
  - UZ Leuven, Leuven
  - C. H. U. Sart-Tilman; Laboratory, Liège
  - CHU UCL Namur / site Godinne, Yvoir
- Canada (5):
  - Synergy Respiratory Care, Sherwood Park, Alberta
  - Kelowna Respiratory and Allergy Clinic, Kelowna, British Columbia
  - The Rhema Research Institute, Owen Sound, Ontario
  - Dr. Syed Anees Medicine Profession Corporation, Windsor, Ontario
  - C.I.C. Mauricie, Trois-Rivières, Quebec
- China (10):
  - Beijing Friendship Hospital Affiliated of Capital University of Medical Science, Beijing
  - Peking Union Medical College Hospital; Pharmacy, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital Of Central South University, Changsha
  - Shengjing Hospital of China Medical University, Shenyang
  - Hebei Medical University - The Second Hospital, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Wuxi People's Hospital, Wuxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni Nemocnice; Interni Klinika - odd. Invazivni Kardiologie, Hradec Králové
  - Thomayerova nemocnice; Lekarna - pavilon H, Prague
  - Krajska nemocnice T. Bati a.s.; Neurologicke oddeleni, Zlín
- Denmark (2):
  - Gentofte Hospital, Hellerup
  - Odense Universitetshospital, Odense C
- France (13):
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Regional Universitaire de Brest - Hopital de la Cavale Blanche, Brest
  - Hopital Louis Pradel, Bron
  - CHU Hopitaux de Bordeaux, CHU Hopitaux de Bordeaux
  - CHU Dijon Bourgogne Hôpital François Mitterand, Dijon
  - CHU de Grenoble - Hôpital André Michallon; Pole Pharmacie, La Tronche
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Servie de Pneumologie et centre de Transplantation Pulmonaire, Marseille
  - CHU Nice - Hôpital Pasteur 2, Nice
  - Hopital Bichat Claude Bernard; Hepatologie Gastro Enterologie, Paris
  - Centre Hospitalier Universitaire de Reims; l'Hopital Maison Blanche, Reims
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - CHU Tours - Hôpital Bretonneau, Tours
- Germany (6):
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Thoraxklinik-Heidelberg gGmbH; Apotheke der Thoraxklinik, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Praxis für Pneumologie Dr. Silke Mronga & Dr. Lukas Jerrentrup, Marburg
  - Lungenklinik Münnerstadt, Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Krankenhaus Bethanien gGmbH, Solingen
- Greece (9):
  - Evangelismos Hospital; Endocrinology, Diabetes & Metabolism, Athens
  - Attikon University General Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklio
  - University Hospital of Ioannina; Pulmonology Department, Ioannina
  - Athens Medical Center, Marousi
  - University of Thessaly Faculty of Medicine, Mezourlo
  - University General Hospital of Patras, Pátrai
  - "General hospital of Chest Diseases ""Sotiria"", 7th Pulmonary Clinic ", Sotiria Athens
  - General Hospital of Thessaloniki G. Papanikolaou, Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital; Dept. of Medicine & Therapeutics, Hong Kong
  - The University of Hong Kong; Queen Mary Hospital, Hong Kong
- Hungary (5):
  - Semmelweis University, Budapest
  - Debreceni Egyetem, Debrecen
  - Markusovszky Egyetemi Oktatokorhaz ; SZEMESZET, Szombathely
  - Szent Borbala Korhaz, Tatabánya
  - Tudogyogyintezet Torokbalint; Onkologiai és Jarobeteg Centrum, Törökbálint
- Israel (12):
  - Barzilai Medical Center; Neurology Department, Ashkelon
  - Ben-Gurion University of the Negev - Soroka University Medical Center - Pulmonology Institute, Beersheba
  - Shamir medical center, Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petach Tiqwa
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center; Department of Neurology, Tel Aviv
- Italy (20):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Abruzzo
  - Policlinico Riuniti di Foggia - Department of Medical and Surgical Sciences - University of Foggia, Foggia, Apulia
  - "AZIENDA OSPEDALIERA DEI COLLI Monaldi-Cotugno-CTO - Pneumologia ", Napoli, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Ospedale Morgagni Pierantoni; Patologia clinica, Forlì, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Policlinico Tor Vergata - U.O.C. Malattie Apparato Respiratorio, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli; Servizio di Farmacia, Rome, Lazio
  - Ospedale San Giuseppe; U.O. di Pneumologia, Milan, Lombardy
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Fondazione IRCCS Policlinico San Matteo Divisione di EmatologiaDipartimento di Onco-Ematologia, Pavia, Lombardy
  - A.O.U. Sassari; Dip. Medicina Clinica e Sperimentale, Sassari, Sardinia
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania, Sicily
  - Az. Osp. Univ. P. Giaccone; UOC di Pneumologia, Palermo, Sicily
  - Ismett Istituto Mediterraneo Trapianti E Terapie Alta Specializzazione;Pneumologia, Palermo, Sicily
  - AOUC Azienda Ospedaliero-Universitaria Careggi; Neurologia 2, Florence, Tuscany
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; Dip. Medicina clinica e Scienze Immunologiche, Siena, Tuscany
  - Azienda Ospedale Universita Di Padova; Divisione Clinicizzata Di Nefrologia 1, Padua, Veneto
  - University of Padova Ca' Foncello Hospital Immunologic & Respiratory Rare Diseases Center, Treviso, Veneto
- Japan (20):
  - Nagoya University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Kobe City Medical Center General Hospital, Hyōgo
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kameda Medical Center, Kamogawa
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kawasaki-Shi
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Ibarakihigashi National Hospital; Center for Clinical Research, Naka-gun
  - Kurashiki Central Hospital, Okayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi
  - Tosei General Hospital, Seto-shi
  - Tenri Hospital, Tenri-Shi
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Tokyo Medical Ando Dentaluni Hospital Faculty of Medicine; Surgical Oncology, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
- Mexico (5):
  - INER- Instituto Nacional de Enfermedades Respiratorias"Ismae, Mexico City, Mexico CITY (federal District)
  - Centro Respiratorio de México, México, Mexico CITY (federal District)
  - Unidad Médica para la Salud Integral UMSI, San Nicolás de los Garza, Nuevo León
  - Unidad de Investigacion CIMA SC, Chihuahua City
  - CICC Morelia, Morelia
- Netherlands (2):
  - Sint Antonius Ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - NZ Respiratory & Sleep Institute, Auckland
  - University of Otago, Christchurch, Christchurch
  - Waikato Hospital; Gastro Research, Hamilton
  - Tauranga Hospital, Tauranga
- Norway (3):
  - Helse Bergen HF Haukeland universitetssykehus; Hudavdelingen, Bergen
  - Akershus universitetssykehus, Lørenskog
  - Oslo University Hospital HF, Rikshospitalet, Oslo
- Poland (3):
  - Centrum Medycyny Oddechowej Mroz sp. j., Bia?ystok
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
- Portugal (4):
  - Hospital de Braga; Centro Clínico Académico (Piso 1, Ala E), Braga
  - Centro Hospitalar do Alto Ave; EPE, Guimarães
  - Centro Hospitalar Universitario Lisboa Norte - Hospital Pulido Valente, Lisbon
  - CHVNG/E_Unidade 1; Servico de Pneumologia, Vila Nova de Gaia
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital; Oncology, Singapore
- South Africa (2):
  - University of Cape Town Lung Institute; Lung Clinical Research, Cape Town
  - Vergelegen Medi-Clinic, Somerset West
- South Korea (9):
  - The Catholic University of Korea Bucheon St. Mary's Hospital, Gyeonggi-do
  - Gacheon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam-si
  - The Catholic University of Korea Yeouido St. Mary's Hospital; Hematology-Oncology, Seoul
  - Seoul National University Hospital (SNUH) - Medical Oncology Center, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (22):
  - HUA - Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitaria Parc Taulí; Servicio de Neurología, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - CHUS H Clinico U de Santiago, Santiago de Compostela, LA Coruña
  - Hospital Universitario del Henares, Coslada, Madrid
  - Hospital Univ. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neumologia, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Virgen de las Nieves; Servicio de Neumologia, Granada
  - Hospital Universitario de la Princesa; Servicio de Aparato Digestivo, Madrid
  - Clinica Universidad de Navarra ; Servicio de Farmacia, Madrid
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario La Paz, Madrid
  - Hospital Ramón y Cajal;Servicio de Neumología, Madrid
  - Fundacion Jimenez Diaz-UTE, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (7):
  - Buddhist Tzu Chi Dalin General Hospital; Rheumatology, Chiayi City
  - Kaohsiung Medical University Hospital; Chung-Ho Memorial Hospital, Kaoshiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Far Eastern Memorial Hospital; Department of Clinical Pathology, Taipei
  - Veterans General Hospital - Taichung, Xitun Dist.
- Turkey (Türkiye) (14):
  - Istanbul Universitesi Onkoloji Enstitüsü Hastanesi, ?stanbul
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi; Balcali, Adana
  - Ankara Universitesi Tip Fakultesi Hastaneleri - Cebeci Hastanesi, Ankara
  - Uludag Universitesi - Saglik Uygulama ve Arastirrma Merkezi, Bursa
  - Gaziantep Universitesi Tip Fakultesi, Gaziantep
  - Yedikule Gogus Hastaliklari ve Gogus Cerrahisi Egitim ve Arastirma Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Dokuz Eylul University Faculty of Medicine; Chest Diseases, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Marmara Universitesi Hastanesi Marmara University Hospital, Maltepe
  - Eriyes universitesi T?p Fakultesi Hastanesi, Melikgazi/Kayser
  - Mersin Universitesi Tip Fakultesi Hastanesi; Tibbi Onkoloji Birimi, Mersin
  - Akdeniz University Faculty of Medicine Department of Pulmonology, Muratpasa/Antalya
  - Koc Universitesi (KU) Tip Fakultesi (Koc University School of Medicine), Sarıyer

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Mantovani A, Garlanda C. Humoral Innate Immunity and Acute-Phase Proteins. N Engl J Med. 2023 Feb 2;388(5):439-452. doi: 10.1056/NEJMra2206346. No abstract available. PMID 36724330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 48 investigative sites in 16 countries.
Groups:
- Cohort A: Zinpentraxin Alfa: Participants entered this Cohort following participation in study PRM-151-202.
- Cohort B: Ex-Placebo; Cohort B: Zinpentraxin Alfa: Participants entered, following participation in study WA42293.
Period: Overall Study
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Started | 21 | 49 | 47
Completed | 0 | 0 | 0
Not Completed | 21 | 49 | 47
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 2 | 2
Not completed — Lung Transplant | 0 | 0 | 1
Not completed — Grade 4 infusion related reaction (IRR) | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 19 | 47 | 41
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa | Total
Number analyzed (Participants) | 21 | 49 | 47 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.5 (5.5) | 74.6 (7.6) | 73.2 (6.8) | 74.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 10 | 25
  Male | 16 | 39 | 37 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 7
  Not Hispanic or Latino | 18 | 47 | 45 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 19 | 47 | 43 | 109
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant who was administered a pharmaceutical product, regardless of causal attribution. Grading was completed according to the CTCAE, version 5.0.
Time Frame: From baseline until 8 weeks after the final dose, an average of 6 months
Population: The safety-evaluable population included all enrolled participants who received at least one administration (full or partial dose) of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Participants | 18 | 25 | 26

2. Primary Outcome: Percentage of Participants With Infusion Related Reactions (IRRs) and Other AEs of Special Interest
Description: IRRs were defined as AEs that occurred during or within 24 hours after study drug administration and were judged to be related to study drug infusion.
Time Frame: From baseline until 8 weeks after the final dose, an average of 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Participants | 2 | 2 | 4

3. Primary Outcome: Percentage of of Participants Permanently Discontinuing Study Treatment Due to AEs
Time Frame: From baseline until 8 weeks after the final dose, an average of 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Participants | 2 | 2 | 1

4. Secondary Outcome: Annual Rate of Change in Forced Vital Capacity (FVC) (mL)
Time Frame: From baseline until study completion (up to approximately 1.5 years)
Population: The full analysis set included all enrolled participants who received at least one administration (full or partial dose) of study drug.
Measure: Mean (95% Confidence Interval); unit: Milliliter (mL)
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Milliliter (mL) | -229.12 [-317.39 to -140.9] | -272.96 [-698.97 to 153.06] | -120.77 [-546.26 to 294.73]

5. Secondary Outcome: Annual Rate of Change in 6-Minute Walk Distance (6MWD)
Time Frame: From baseline until study completion (up to approximately 1.5 years)
Population: The full analysis set included all randomized participants who received at least one administration (full or partial dose) of study drug and used the grouping according to the treatment assignment at randomization.
Measure: Mean (95% Confidence Interval); unit: Meters (m)
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Meters (m) | -86.95 [-170.80 to -3.10] | 64.64 [-98.62 to 227.90] | -163.66 [-324.02 to -3.30]

6. Secondary Outcome: Annual Rate of Change in FVC% Predicted
Time Frame: From baseline until study completion (up to approximately 1.5 years)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Percent predicted
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Percent predicted | -6.96 [-9.70 to -4.22] | -6.91 [-14.77 to 0.96] | -3.37 [-11.18 to 4.44]

7. Secondary Outcome: Change in Carbon Monoxide Diffusing Capacity (DLCO)
Time Frame: At Baseline, Week 24 and Week 48
Population: The full analysis set included all randomized participants who received at least one administration (full or partial dose) of study drug and used the grouping according to the treatment assignment at randomization. In the Ex-placebo arm, no participant was assessed for DLCO after baseline. Due to short length of follow-up, no DLCO assessment was collected at Week 48 for Cohort B: Zinpentraxin Alfa arm.
Measure: Mean (Standard Deviation); unit: DLCO% Predicted
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 11 | 36 | 28
DLCO% Predicted
  Baseline | 40.20 (16.29) | 44.91 (10.94) | 42.27 (11.14)
  Week 24: number analyzed (Participants) | 5 | 0 | 1
  Week 24 | 1.08 (4.05) |  | -1.55 (NA) — Cannot take the standard deviation from one participant.
  Week 48: number analyzed (Participants) | 5 | 0 | 0
  Week 48 | -2.80 (3.76) |  |

8. Secondary Outcome: Time to Disease Progression
Description: Time to first occurrence of >=10% absolute decline in % predicted FVC, >=15% relative decline in 6MWD, or death
Time Frame: From baseline until study completion (up to approximately 1.5 years)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Months | 5.6 [2.9 to 8.3] | NA [NA to NA] — Due to the low number of events and early termination of the study, the median and 95% CI weren't estimable. | NA [NA to NA] — Due to the low number of events and early termination of the study, the median and 95% CI weren't estimable.

9. Secondary Outcome: Survival
Time Frame: Every 6 Months and at study completion (up to approximately 1.5 years)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Months | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable. | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable. | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable.

10. Secondary Outcome: IPF-related Mortality
Time Frame: Every 6 Months and at study completion (up to approximately 1.5 years)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Months | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable. | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable. | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable.

11. Secondary Outcome: Respiratory-related Mortality
Time Frame: Every 6 Months and at study completion (up to approximately 1.5 years)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 49 | 47
Months | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable. | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable. | NA [NA to NA] — Due to the low number of events, the median and 95% CI was not estimable.

12. Secondary Outcome: Plasma Concentrations of PRM-151 at Specified Timepoints
Description: Due to early termination of the study, only participants enrolled in Cohort A receiving at least one IV dose of zinpentraxin alfa had their plasma concentrations analyzed.
Time Frame: Days 1 and 5, Weeks 4, and 12
Population: The pharmacokinetic population included all randomized participants who received at least one administration (full or partial dose) of zinpentraxin alfa and at least one evaluable postdose PK sample that was above the lower limit of quantification (LLOQ).
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 21 | 0
micrograms per millilitre (ug/mL)
  Day 1 -pre infusion: number analyzed (Participants) | 0 | 0
  Day 1 - 2h Post Infusion: number analyzed (Participants) | 20 | 0
  Day 1 - 2h Post Infusion | 203.85 (55.72) |
  Day 5 - Pre Infusion | 42.83 (18.89) |
  Day 5 - 2h Post Infusion: number analyzed (Participants) | 20 | 0
  Day 5 - 2h Post Infusion | 252.90 (53.42) |
  Week 4 - Pre Infusion: number analyzed (Participants) | 18 | 0
  Week 4 - Pre Infusion | 2.50 (0) |
  Week 4 - 2h Post Infusion: number analyzed (Participants) | 18 | 0
  Week 4 - 2h Post Infusion | 209.00 (42.93) |
  Week 12 - Pre Infusion: number analyzed (Participants) | 17 | 0
  Week 12 - Pre Infusion | 2.50 (0.00) |
  Week 12 - 2h Post Infusion: number analyzed (Participants) | 17 | 0
  Week 12 - 2h Post Infusion | 215.65 (50.47) |

13. Secondary Outcome: Prevalence of Anti-drug Antibodies (ADAs) to PRM-151 at Baseline
Description: Due to early termination of the study, only ADA samples from participants in Cohort A were analyzed.
Time Frame: Baseline (Day 1)
Population: The immunogenicity population included all randomized participants with at least one postdose ADA assessment and were grouped according to treatment received or, if no treatment is received prior to study discontinuation, according to treatment assigned.
Measure: Number; unit: Participants
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B: Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 20 | 0 | 0
Participants | 0 |  |

14. Secondary Outcome: Percentage of Participants With ADAs During the Study
Description: Due to early termination of the study, only ADA samples from participants in Cohort A were analyzed.
Time Frame: Weeks 4, 12 and 24
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Groups:
- Cohort B Ex-Placebo; Cohort B: Zinpentraxin Alfa: Participants entered, following participation in study WA42293.
Arm/Group | Cohort A: Zinpentraxin Alfa | Cohort B Ex-Placebo | Cohort B: Zinpentraxin Alfa
Number analyzed (Participants) | 20 | 0 | 0
Percentage of Participants | 0 |  |

ADVERSE EVENTS:
Time Frame: AEs were assessed from baseline until 8 weeks after the final dose, an average of 6 months. Deaths were assessed for up to 1.5 years.
Groups:
- Cohort A Zinpentraxin Alfa: Participants entered this Cohort following participation in study PRM-151-202.
- Cohort B Zinpentraxin Alfa: Participants entered, following participation in study WA42293.
Arm/Group | Cohort A Zinpentraxin Alfa | Cohort B Ex-Placebo | Cohort B Zinpentraxin Alfa
All-Cause Mortality (participants affected / at risk) | 0/21 | 2/49 | 2/47
Serious Adverse Events (participants affected / at risk) | 5/21 | 8/49 | 6/47
Other Adverse Events (participants affected / at risk) | 14/21 | 16/49 | 14/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Zinpentraxin Alfa (N=21) | Cohort B Ex-Placebo (N=49) | Cohort B Zinpentraxin Alfa (N=47)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Zinpentraxin Alfa (N=21) | Cohort B Ex-Placebo (N=49) | Cohort B Zinpentraxin Alfa (N=47)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (4)
Fatigue (General disorders) | 2 (3) | 3 (3) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4) | 6 (6) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 2 (4) | 4 (4)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to the Sponsor's decision to terminate the parent study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04594707/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04594707/SAP_001.pdf